CLINICAL TRIAL: NCT07044453
Title: Risk-adapted Adjuvant Chemotherapy Guided by the Tumour Stage for Operated Pancreatic Adenocarcinoma Following Neoadjuvant Chemotherapy With mFOLFIRINOX - A Multicenter, FRENCH-PRODIGE Randomized Comparative Phase II/III Trial FRENCH26 - PRODIGE93 - PANACHE 02 Trial
Brief Title: Risk-adapted Adjuvant Chemotherapy Guided by the Tumour Stage for Operated Pancreatic Adenocarcinoma Following Neoadjuvant Chemotherapy With mFOLFIRINOX
Acronym: PANACHE 02
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Partenariat de Recherche en Oncologie DIGEstive - PRODIGE (Unknown); Federation de recherche en chirurgie digestive (FRENCH) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021/0377/HP; 2024-519048-33-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-13; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Resected Pancreatic Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group - Arm A: (Experimental): Adjuvant chemotherapy guided by pathological analysis (downstaging)
  * pT1-2/N0/R0 status: 3 months mFOLFIRINOX adjuvant chemotherapy (no change in chemotherapy regimen compared to neoadjuvant setting)
  * pT3-4 or N+ or R1 status: 3 months Gemcitabine with NabPaclitaxel adjuvant chemotherapy (change in chemotherapy regimen compared to neoadjuvant setting).
  Interventions: Drug: Gem/Nabpaclitaxel infusion; Drug: mFOLFIRINOX infusion
- Control group - Arm B (Active Comparator): 3 months mFOLFIRINOX adjuvant chemotherapy regardless of pathological analysis
  Interventions: Drug: mFOLFIRINOX infusion

INTERVENTIONS:
Drug: Gem/Nabpaclitaxel infusion — Downstaging and pathological response is empirically define as T1-2/N0/R0 status. If the anatomopathological analysis shows a lesion classified as T3-4 or N+ or R1, an adjuvant chemotherapy based on Gemcitabine with Nab Paclitaxel will be proposed for a period of 3 months.
  Arms: Experimental group - Arm A:
Drug: mFOLFIRINOX infusion — Downstaging and pathological response is empirically define as T1-2/N0/R0 status. In that setting the patients will receive mFOLFIRINOX adjuvant chemotherapy 3 months.

SUMMARY:
Induction mFOLFIRINOX has become the standard in the management of locally advanced and borderline adenocarcinoma. Following the results of the PREOPANC-01 JASP-05, NEONAX studies it is expected that the neoadjuvant approach will be the standard strategy soon in patients with resectable PAC. The results of the PANACHE-01 trial confirm the feasibility of the neoadjuvant approach in the setting of resectable adenocarcinoma. Two randomized phase III studies, on the same design as PANACHE-01 are currently underway comparing neoadjuvant and adjuvant chemotherapy with mFOLFIRINOX for resectable PAC, (Alliance AO21806, NCT04340141; PREOPANC3, NCT04927780). Despite the improvement of oncosurgical management, recurrence of PAC soon after resection occurs frequently, leading to the dismal prognosis and unnecessary surgery-related loss of quality of life. Thus, there is urgent need for development of innovative and new strategies to decrease postoperative recurrence.

Important residual tumor load after NAT suggests a primary resistance of the tumor or the selection of resistant clones. The most innovative aspect of this study will be to adapt the adjuvant chemotherapy strategy to the pathological response (downstaging) in patients who will have R0-R1 resection after neoadjuvant mFOLFIRINOX, taking into account the chemoresistance/sensibility status of the tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed resected pancreatic adenocarcinoma (R0 or R1) who received 3 months of neoadjuvant mFOLFIRINOX, including anatomically resectable and borderline resectable tumors, in accordance with the definitions and therapeutic considerations provided in the TNCD (2024), and ESMO (2023) guidelines.
2. Performans status ECOG 0 or 1
3. CA 19-9 level ≤ 200 U/ml
4. Age 18 or over
5. Absolute neutrophil count > 1,500 mm3 platelet count > 100,000 mm3 creatinine clearance (according MDRD equation) > 50 ml/min, haemoglobin level > 10 g/dl (transfusions are authorized)
6. Women of childbearing potential (a woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile):

   * with highly effective contraception (Cf. CTCG) combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomised partner, sexual abstinence) since 1 month, during chemotherapy treatment and for 15 months after cessation of chemotherapy treatment and,
   * a negative blood pregnancy test by B-HCG at inclusion as well as pregnancy tests before each cycle of adjuvant chemotherapy, then monthly throughout the study until 15 months after the end of exposure to systemic treatment
   * Women permanently sterile (hysterectomy, bilateral salpingectomy and bilateral oophorectomy)
   * Postmenopausal women: A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
7. For men participating in the study, contraception is required during the trial and for 12 months after stopping chemotherapy treatment.
8. Patient affiliated with, or beneficiary of a social security (national health insurance) plan
9. Patient able to comply with the study protocol, in the investigator's judgment
10. Read and understood the information letter and signed the consent form

Exclusion Criteria:

1. Metastatic PAC on post-operative imaging
2. Cholangiocarcinoma, ampullary carcinoma or other Non PAC pancreatic tumors
3. Non-controlled congestive heart failure - non-treated angina; recent myocardial infarction (In the previous year) - non-controlled AHT (SBP >160 mm or DBP > 100 mm, despite optimal drug treatment), long QT
4. Major non-controlled infection, chronic infectious diseases, immune deficiency syndromes
5. Premalignant hematologic disorders, e.g. myelodysplastic syndrome
6. Severe liver failure
7. Past or current history of malignancies except for the indication under this study and curatively treated Basal and squamous cell carcinoma of the skin, In-situ carcinoma of the cervix, Other malignant disease without recurrence after at least 2 years of follow-up
8. Any medical, psychological or social situation that (in the investigator's opinion) could limit the patient's compliance with the protocol or the ability to obtain or interpret data or to understand the conditions required for his/her participation to the protocol or unable him/her to give an informed consent
9. Pregnant or breastfeeding women and women of child-bearing age not using effective means of contraception
10. Person participating to another interventional research having the same primary endpoint
11. Person deprived of liberty by an administrative or judiciary decision or person placed under judicial protection, under guardianship or curatorship
12. Uracilemia ≥ 150 ng/ml (suggestive of complete DPD deficiency)
13. Contraindication to study adjuvant chemotherapy treatments in accordance with the SmPC's of the products used in this trial (Gemcitabine, Nab-Paclitaxel, Oxaliplatin, Folinic Acid or Leucovorin, Irinotecan, Fluorouracil) -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | from enrollment up to 5 years
  The primary efficacy endpoint is the Disease Free Survival at 2 years (DFS), defined as the time from randomization to locoregional recurrence, occurrence of distant metastases or second pancreatic cancer, or death (all causes) whichever occurred first. Patients free of events will be censored at the date of the last disease evaluation either during study treatment period or during follow-up period
Overall Survival | from enrollment up to 7 years
  The primary efficacy endpoint is the Overall Survival at 3 years(OS), defined as the time from randomization to the death from any cause. Alive patient will be censored at last date known to be alive either during study treatment period or during follow-up period

SECONDARY OUTCOMES:
Incidence and grade for Adverse Events (AEs) | from enrollment up to 7 years
  drug related AEs, drug related AE leading to dose reduction or discontinuation during treatment, SAE and SUSAR, according to NCI-CTCAE V5.0.
metastatic recurrence free survival in both arms | from enrollment up to 7 years
  Time to metastatic recurrence defined as the time from randomization to occurrence of distant metastases.
rate of patients with early recurrence | from enrollment up to 5 years
  Early recurrence < 6 months after surgical randomization
evolution of the health-related quality of life | from enrollment up to 7 years
  Health related quality of life EORTC QLQ-C30 and QLQ-PAN26 questionnaires
Correlation of tumour response with TNM classification | from enrollment up to 7 years
  TNM classification :
  T- the extent of the primary tumour (T1-T4 Increasing size) N- the absence N0 or presence (N1-N2) and extent of regional lymph node metastasis M- the absence (M0) or presence (M1) of distant metastasis
Correlation of tumour response with Residual Tumour (R) Classification | from enrollment up to 7 years
  Residual Tumour (R) Classification : R0 No residual tumour R1 Microscopic residual tumour

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: Undecided